CLINICAL TRIAL: NCT01012921
Title: Straumann® MembraGel Comparison of a PEG Membrane and a Collagen Membrane for the Treatment of Bone Dehiscence Defects at Bone Level Implants
Brief Title: Comparison of a PEG Membrane and a Collagen Membrane for the Treatment of Bone Dehiscence Defects at Bone Level Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 07/07
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-05

CONDITIONS: Degeneration; Bone
Keywords: GBR; GTR; Dental Implant surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bio-Gide® membrane (Active Comparator): Bio-Gide® membrane This is a biodegradable bilayer membrane for bone and tissue regeneration. It has a natural collagen structure and is of porcine origin
  Interventions: Device: barrier membrane; Other: Bio-Gide® membrane
- MembraGel (Experimental): MembraGel The Straumann membrane is a synthetic degradable barrier membrane
  Interventions: Device: barrier membrane; Device: MembraGel

INTERVENTIONS:
Device: barrier membrane — The in situ forming gel serves as a barrier membrane for Guided Bone Regeneration (GBR).
Device: MembraGel — Device application at surgery
  Other Names: Straumann® MembraGel
  Arms: MembraGel
Other: Bio-Gide® membrane — Device application at surgery
  Arms: Bio-Gide® membrane

SUMMARY:
The aim of the study is to test in a randomized comparative study the performance of Straumann® MembraGel (PEG Membrane) to act as a barrier for guided bone regeneration compared to that of a standard collagen membrane (BioGide®) in the bone regeneration around Straumann® SLActive bone level titanium implants.

Furthermore the clinical evaluation and comparison of complementary parameters describing the bony and soft tissue environments at the surgical sites during the study period to evaluate effectiveness and performance of the membranes.

DETAILED DESCRIPTION:
At the primary endpoint of the study - 6 month post-operative - the vertical bone gain will be measured for changes.

The changes will be evaluated by measuring the distance between the implant shoulder and the first visible bone contact on the implant. The measurement will be taken on the medial and distal aspect on the implant at site of interest. Measurements will take into account distortion based on changes on the radiograph from the true dimension of the implant.

Intra-oral photographs will be taken at each study visit to document the initial appearance of the soft tissue and the subsequent healing of the soft tissue post-implant placement. The photographs will be taken buccal and occlusial at study site of interest.

The physical appearance of soft tissue (form, colour, tissue biotype, surface aspect) will be clinically assessed by visual inspection.

In addition changes in the high of the keratinized gingiva will be assessed in mm. This will be measured mid-crestal in buccal direction to the mucogingival border by a periodontal probe.

Changes in gingival recession will be measured at the implant leading visit and the yearly follow-up visit 18, 30 and 42 month post surgery. The distance between the margin of the gingiva and the edge of the crown will be assessed at accessible buccal, palatal, distal and medial sites.

A measurement of vertical defect height will be performed evaluating the distance of the implant shoulder to the first bone to implant contact at surgery visit and 6-month later.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntarily signed the informed consent form before any study related action
* Males and females must be at least 18 years of age and not more than 80 year old.
* Have at least one missing tooth in the posterior mandible or maxilla in quadrant 1, 2, 3, 4 (FDI positions 4-7), requiring one or more dental implants.
* Partially edentulous patients and patients in need of a fixed dental prosthesis
* The tooth at the implant site(s) must have been extracted or lost at least 6 weeks before the date of implantation.
* Bone defect(s) must be present with a vertical dimension greater than or equal to 3 mm at the foreseen GBR site measured after dental implant placement.
* Full mouth bleeding on Probing (FMBoP) and full mouth plaque score (FMPI) are both lower or equal than 25%
* Patients must be committed to the study.

Exclusion Criteria:

* Presence of conditions requiring chronic routine prophylactic use of antibiotics (e.g., history of rheumatic heart disease, bacterial endocarditis, cardiac valvular anomalies, prosthetic joint replacements)
* Major systemic diseases
* Medical conditions requiring prolonged use of steroids
* Use of Bisphosphonate intravenously
* Current pregnancy or breastfeeding women
* Physical or mental handicaps that would interfere with the ability to perform adequate oral hygiene
* Alcoholism or chronically drug abuse
* Immunocompromised patients
* Patients who smoke more than 10 cigarettes per day or cigar equivalents, or who chew tobacco
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability.

Local exclusion criteria

* Local inflammation, including untreated periodontitis
* Regenerative treatment necessary adjacent to the planned study site of interest
* Mucosal diseases or oral lesions
* History of local irradiation therapy
* Severe bruxing or clenching habits
* Persistent intraoral infection
* Patients with inadequate oral hygiene or unmotivated for adequate home care
* Previous GBR or GTR treatment at the implant site
* Lack of primary stability of the dental implant at site of interest. In this instance the patient must be withdrawn and the patient treated accordingly (exclusion criteria at surgery)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Haemmerle, Prof. Dr., Principal Investigator — Medical University Zürich, Switzerland
Locations (9):
- Catholic University Leuven School of Dentistry, Oral Pathology & Maxillo-facial Surgery, Leuven, Belgium
- Germany (2):
  - Charite, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
- Semmelweis University, Budapest, Hungary
- Eastman Hospital, Rome, Italy
- Spain (2):
  - Prof. Mariano Sanz, Madrid
  - Clinica Blanco Ramos, Santiago de Compostela
- Gävle Hospital, Gävle, Sweden
- Medical University Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bio-Gide® Membrane | MembraGel
Started | 57 | 60
Completed | 47 | 47
Not Completed | 10 | 13

BASELINE CHARACTERISTICS:
Population: Analysis population is PP
Groups:
- Total: Total of all reporting groups
Arm/Group | Bio-Gide® Membrane | MembraGel | Total
Number analyzed (Participants) | 45 | 40 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (14.7) | 50.6 (14.0) | 49.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 33 | 58
  Male | 20 | 7 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 44 | 40 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 3 | 4 | 7
  Belgium | 3 | 2 | 5
  Italy | 8 | 5 | 13
  Switzerland | 5 | 5 | 10
  Germany | 15 | 16 | 31
  Spain | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: The Bone Fill Was Assessed at 6 Months After Regenerative Therapy.
Description: Change between baseline (regenerative therapy) and the 6 months timepoint is reported.
Time Frame: Assessed at 6 months reported
Population: PP
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bio-Gide® Membrane | MembraGel
Number analyzed (Participants) | 45 | 40
mm | 3.2 (2.1) | 2.5 (1.5)

ADVERSE EVENTS:
Arm/Group | Bio-Gide® Membrane | MembraGel
Serious Adverse Events (participants affected / at risk) | 0/57 | 1/60
Other Adverse Events (participants affected / at risk) | 6/57 | 18/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bio-Gide® Membrane (N=57) | MembraGel (N=60)
Cerebral hemorrhagic infarction (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bio-Gide® Membrane (N=57) | MembraGel (N=60)
Infection (Infections and infestations) | 2 | 10
Delayed epithelisation (Infections and infestations) | 1 | 2
Swelling (Infections and infestations) | 1 | 2
Allergy (Immune system disorders) | 1 | 1
Dehiscence (General disorders) | 1 | 1
Lack of osseointegration (General disorders) | 0 | 2
Pain (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No